CLINICAL TRIAL: NCT01492010
Title: Role of Leucine in the Regulation of Human Myofibrillar Protein Synthesis at Rest and Following Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of California, Davis (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEU-10-141
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Regulation of Muscle Protein Synthesis
Keywords: skeletal muscle; FSR; resistance exercise; leucine; protein
MeSH Terms: interventions — Whey Proteins; Leucine; Amino Acids, Essential

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25 g protein (Experimental): 25 g whey protein
  Interventions: Dietary Supplement: whey protein
- 6.25 g protein supplemented with leucine (Experimental): 6.25 g protein supplemented with leucine
  Interventions: Dietary Supplement: whey protein supplemented with leucine
- 6.25 g whey protein with EAA (Experimental): 6.25 g protein supplemented with a mixture of essential amino acids devoid of leucine
  Interventions: Dietary Supplement: whey protein supplemented with essential amino acids

INTERVENTIONS:
Dietary Supplement: whey protein — 25 g whey protein
  Other Names: whey protein powder
  Arms: 25 g protein
Dietary Supplement: whey protein supplemented with leucine — 6.25 g whey protein supplemented with free form leucine
  Other Names: whey protein powder supplemented with free-form leucine
  Arms: 6.25 g protein supplemented with leucine
Dietary Supplement: whey protein supplemented with essential amino acids — 6.25 g whey protein supplemented with essential amino acids devoid of leucine
  Other Names: whey protein supplemented with EAA devoid of leucine
  Arms: 6.25 g whey protein with EAA

SUMMARY:
Muscle mass is normally maintained through the regulated balance between the processes of protein synthesis (i.e. making new muscle proteins) and protein breakdown (breaking down old muscle proteins). Proteins are composed of amino acids and we know that amino acids increase muscle protein synthesis. However, not all amino acids are the same. Essential amino acids are ones that must be consumed through food, while non-essential amino acids can be made by our body. Interestingly, the essential amino acids are all that are required to increase the rate of muscle protein synthesis. In addition, the essential amino acid leucine appears to be particularly important in regulating protein synthesis. However, how leucine is able to increase protein synthesis is not entirely understood. Previously, it has been shown that 20-25 g of high-quality protein, such as that found in milk, appears to be the amount of protein that maximizes the rate of muscle protein synthesis after performing a bout of resistance exercise. Thus, the aim is to measure the synthesis of new muscle proteins after ingesting the following:

1. 25g whey protein
2. 6.25g whey protein supplemented with leucine
3. 6.25g whey protein supplemented with essential amino acids but no leucine

The investigators will measure muscle protein synthesis after consumption of the above beverages in a leg that has done no exercise ( ie. a rested leg) and in the other leg that has done resistance exercise. The hypothesis is that 6.25g whey supplemented with leucine will stimulate muscle protein synthesis as effectively as 25g whey, but that 6.25g whey supplemented will all the essential amino acids except whey will be less effective at increasing muscle protein synthesis. Whey protein is a dairy-based protein found in cow's milk, thus when you drink a glass of milk you are consuming some whey protein. However, the investigators will be using an isolated form of whey protein, meaning it has been removed from milk. As mentioned previously, amino acids are 'strung-together' to make protein. The 'essential' amino acids must be consumed through food because our body cannot make them, thus they are consumed when you eat protein-rich foods like milk or chicken.

ELIGIBILITY:
Inclusion Criteria:

* male
* 18-35 years of age
* non-smoker/ non-tobacco product user

Exclusion Criteria:

* heart disease
* vascular disease
* rheumatoid arthritis
* diabetes
* poor lung function
* uncontrolled blood pressure
* dizziness
* thyroid problems

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 5 hours postprandial
  Muscle protein synthesis will be expressed as fractional synthetic rate (FSR) by dividing the increment in enrichment in the product, i.e. protein-bound C13phe, by the enrichment of the precursor (= intracellular availability).

SECONDARY OUTCOMES:
Signaling molecule phosphorylation status | 1, 3, and 5 hours
  Western blot will be used to measure the phosphorylation status of signaling molecules involved in protein synthesis ie. mTOR, p70S6k, 4E-BP1.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Churchward-Venne TA, Burd NA, Mitchell CJ, West DW, Philp A, Marcotte GR, Baker SK, Baar K, Phillips SM. Supplementation of a suboptimal protein dose with leucine or essential amino acids: effects on myofibrillar protein synthesis at rest and following resistance exercise in men. J Physiol. 2012 Jun 1;590(11):2751-65. doi: 10.1113/jphysiol.2012.228833. Epub 2012 Mar 25. PMID 22451437